CLINICAL TRIAL: NCT02591576
Title: Long Term Excess Mortality of Acute Myocardial Infarction in Patients With and Without Diabetes: A Population-based Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Oras Alabas, Dr, University of Leeds
Other Study IDs: NIGB: ECC 1-06 (d)/2011
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Effect of Diabetes on Long Term Excess Mortality Following Acute Myocardial Infarction
Keywords: Diabetes; ST-elevation myocardial infarction (STEMI); non-STEMI; Excess mortality; Relative survival
MeSH Terms: conditions — Diabetes Mellitus; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ST-elevation myocardial infarction (STEMI)
- non-ST-elevation myocardial infarction (NSTEMI)

SUMMARY:
Diabetes is key risk factor for death following acute myocardial infarction. However, the long-term excess risk of death associated with diabetes following acute myocardial infarction not known. Investigators aimed to determine the long-term excess risk of death associated with diabetes among patients with ST-elevation myocardial infarction (STEMI) and non-STEMI (NSTEMI) after adjustment for multimorbidity, risk factors and cardiac treatments.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Both sex
* 18 years

Exclusion Criteria:

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI and NSTEMI were eligible for analysis if they have been hospitalised following AMI between the period of 2003-2013 and were aged at least 18 years. Only records of the first admission were considered for analyses.
Sampling Method: Non-Probability Sample
Enrollment: 700000 (Actual)
Dates: Start 2003-01; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Long term excess mortality | 8 years

REFERENCES:
- [Derived] Alabas OA, Hall M, Dondo TB, Rutherford MJ, Timmis AD, Batin PD, Deanfield JE, Hemingway H, Gale CP. Long-term excess mortality associated with diabetes following acute myocardial infarction: a population-based cohort study. J Epidemiol Community Health. 2017 Jan;71(1):25-32. doi: 10.1136/jech-2016-207402. Epub 2016 Jun 15. PMID 27307468